CLINICAL TRIAL: NCT03031730
Title: A Phase 1 Dose-Escalation and Exploratory Dose Expansion Study of KRT-232 (AMG 232) in Combination With Carfilzomib, Lenalidomide, and Dexamethasone in Relapsed and/or Refractory Myeloma
Brief Title: Testing the Addition of KRT-232 (AMG 232) to Usual Chemotherapy for Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00099; NCI-2017-00099 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI10076; 10076 (Other: University of Texas MD Anderson Cancer Center LAO); 10076 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2017-01-25; First posted 2017-01-26 (Estimated); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Plasmacytoma; Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Plasmacytoma; Multiple Myeloma | interventions — Specimen Handling; Biopsy; carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AMG 232, carfilzomib, lenalidomide, dexamethasone) (Experimental): Patients receive MDM2 Inhibitor KRT-232 PO QD on days 1-7, carfilzomib IV over 10-30 minutes on days 1-2, 8-9, and 15-16 of cycles 1-12 and on days 1-2 and 15-16 of cycles 13-18, lenalidomide PO on days 1-21, and dexamethasone PO or dexamethasone sodium phosphate IV on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unexpected toxicity. Patients undergo echocardiography during screening and bone marrow biopsy and aspiration, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone Sodium Phosphate; Procedure: Echocardiography; Drug: Lenalidomide; Drug: Navtemadlin

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Carfilzomib — Given IV
  Other Names: Carfilnat; CFZ; Kyprolis; PR 171; PR-171; PR171
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Dexamethasone Sodium Phosphate — Given IV
  Other Names: Cebedex; Corson; Dalalone; Decaject; Dekasol LA; Dexacen; Dexamethasone Sodium Phosphates; Dexasone; Dezone; ReadySharp Dexamethasone; Soludecadron; Solurex; Topidex
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Drug: Navtemadlin — Given PO
  Other Names: (3R,5R,6S)-5-(3-Chlorophenyl)-6-(4-chlorophenyl)-3-methyl-1-((1S)-2-methyl-1-(((1-methylethyl)sulfonyl)methyl)propyl)-2-oxo-3-piperidineacetic Acid; AMG 232; AMG-232; KRT 232; KRT-232; KRT232; MDM2 Inhibitor KRT-232

SUMMARY:
This phase I trial studies the side effects and best dose of MDM2 Inhibitor KRT-232 when given together with carfilzomib, lenalidomide, and dexamethasone in treating patient with multiple myeloma that has come back (relapsed) or has not responded to previous treatment (refractory). KRT-232 (AMG 232) may stop the growth of cancer cells by blocking a protein called MDM2 that is needed for cell growth. Lenalidomide help shrink or slow the growth of multiple myeloma. Drugs used in chemotherapy, such as carfilzomib and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving MDM2 Inhibitor KRT-232, lenalidomide, carfilzomib, and dexamethasone together may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate safety and tolerability of MDM2 Inhibitor KRT-232 (KRT-232 [AMG 232]) in combination with carfilzomib, lenalidomide, and dexamethasone (KRd). (Part A) II. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of KRT-232 (AMG 232) in combination with carfilzomib, lenalidomide, and dexamethasone (KRd). (Part A) III. Confirm the safety and tolerability of KRT-232 (AMG 232) in combination with carfilzomib, lenalidomide, and dexamethasone (KRd) at MTD/tentative RP2D in a goal of 10 subjects with relapsed and/or refractory myeloma. (Part B)

SECONDARY OBJECTIVES:

I. Evaluate pharmacodynamic (PD) effects of KRT-232 (AMG 232) through serum MIC-1 levels. (Part A) II. Assess KRT-232 (AMG 232) exposure-response relationships (PD, toxicity, and efficacy). (Part A) III. Evaluate the overall response rate of KRT-232 (AMG 232) in combination with carfilzomib, lenalidomide, and dexamethasone (KRd) in relapsed/refractory myeloma by International Myeloma Working Group (IMWG) criteria. (Part B) IV. Evaluate PD effects of KRT-232 (AMG 232) through serum MIC-1 levels. (Part B) V. Assess KRT-232 (AMG 232) exposure-response relationships (PD, toxicity, and efficacy). (Part B)

EXPLORATORY OBJECTIVES:

I. To observe and record anti-tumor activity of KRT-232 (AMG 232) in combination with carfilzomib, lenalidomide, and dexamethasone (KRd) in relapsed/refractory myeloma by International Myeloma Working Group (IMWG) criteria. (Part A) II. Evaluate ribonucleic acid (RNA) expression levels of relevant genes in the TP53 pathway that may predict response to therapy using pre- and post-treatment bone marrow biopsies. (Parts A and B)

OUTLINE: This is a dose-escalation study of MDM2 Inhibitor KRT-232.

Patients receive MDM2 Inhibitor KRT-232 orally (PO) once daily (QD) on days 1-7, carfilzomib intravenously (IV) over 10-30 minutes on days 1-2, 8-9, and 15-16 of cycles 1-12 and on days 1-2 and 15-16 of cycles 13-18, lenalidomide PO on days 1-21, and dexamethasone PO or dexamethasone sodium phosphate IV on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unexpected toxicity. Patients undergo echocardiography during screening and bone marrow biopsy and aspiration, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed diagnosis of multiple myeloma
* Subjects must have measurable disease, as defined by at least one of the following:

  * Serum monoclonal protein M-protein level >= 0.5 g/dL
  * Urinary M-protein excretion of >= 200 mg over a 24-hour period
  * Involved free light chain level >= 10 mg/dL, along with an abnormal free light chain ratio
* Subjects must have disease that has relapsed and/or refractory after their most recent therapy, with progressive disease (PD) being defined as an increase of 25% from the lowest response value in any one or more of the following:

  * Serum M-component protein (the absolute increase must be >= 0.5 g/dL) and/or
  * Urine M-component protein (the absolute increase must be >= 200 mg/24 hours) and/or
  * Only in subjects without a measurable serum and urine M protein level: the difference between involved and uninvolved free light chain (FLC) levels (absolute increase) must be > 10 mg/dL
  * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  * Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL) that can be attributed solely to the plasma cell proliferative disorder
* Subjects with one to three lines of therapy for their disease with a line of therapy defined as one or more cycles of a planned treatment program; using this definition, treatment with induction therapy, followed by high dose chemotherapy and autologous stem cell transplantation, and finally by maintenance therapy, would constitute one line, provided that multiple myeloma did not meet criteria for progression at any time during this period
* Subjects must have completed their most recent drug therapy directed at multiple myeloma in the following timeframes:

  * Antitumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, retinoid therapy, hormonal therapy, or investigational agent) at least 21 days prior to cycle 1 day 1 (C1D1) KRT-232 (AMG 232) + KRd
  * Corticosteroids at least 3 weeks prior to starting KRT-232 (AMG 232) + KRd, except for a dose equivalent to dexamethasone of =< 4 mg/day
  * Autologous stem cell transplantation at least 12 weeks prior to starting KRT-232 (AMG 232) + KRd
  * Allogeneic stem cell transplantation at least 24 weeks prior to starting KRT-232 (AMG 232) + KRd, and these subjects must also NOT have moderate to severe active acute or chronic graft versus host disease (GVHD)
* Subjects must be >= 18 years old. Because no dosing or adverse event data are currently available on the use of KRT-232 (AMG 232) in combination with KRd, subjects < 18 years of age are excluded from this study
* Subjects must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,000/mcL without growth factors within 2 week of initiation of treatment
* Platelets >= 50,000 cells/mm^3 if marrow plasmacytosis < 50% OR platelet count >= 30,000 cells/mm^3 if marrow plasmacytosis >= 50%
* Hemoglobin >= 8 g/dL within 2 weeks of the initiation of treatment
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (< 2.0 x ULN for subjects with documented Gilbert's syndrome or < 3.0 x ULN for subjects for whom the indirect bilirubin level suggests an extrahepatic source of elevation)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Alkaline phosphatase < 2.0 x ULN (if liver or bone disease are present, < 3.0 x ULN)
* Creatinine clearance (estimated glomerular filtration rate [eGFR]) >= 50 mL/min/1.73 m^2
* Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN), OR international normalized ratio (INR) < 1.5
* Subjects who have received radiation therapy targeting > 10% of the bone marrow space must have completed this at least 2 weeks prior to starting therapy with KRT-232 (AMG 232) + KRd
* Subjects must be able and willing to provide bone marrow biopsies/aspirates and buccal swab as requested by the protocol
* Subjects must be willing to undergo myeloma genotyping for TP53 mutation, insertion, or deletion at screening
* Subjects must have an estimated life expectancy of at least 3 months
* The effects of KRT-232 (AMG 232) on the developing human fetus are unknown; for this reason and because lenalidomide is known to be teratogenic, women of child-bearing potential must commit to either abstaining continuously from heterosexual sexual intercourse or agree to use 2 forms of adequate contraception or continuously abstain from the time of informed consent for the duration of study participation through 5 weeks (women) after receiving the last dose of KRT-232 (AMG 232), lenalidomide, or carfilzomib; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of KRT-232 (AMG 232) administration; this includes one highly effective form of contraception (e.g. intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (e.g. male latex or synthetic condom, diaphragm, or cervical cap)
* Subjects must be able to swallow medication
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with myeloma that is relapsed and/or refractory to KRd when used in combination defined as progression of disease while on therapy or within 60 days of completing therapy
* Subjects must show evidence of wild-type (WT) p53 status on somatic tissue specimens as assessed by deoxyribonucleic acid (DNA) sequencing; note that since patients with relapsed myeloma have a rapidly proliferating disease, patient can be enrolled and begin treatment prior to obtaining the results of this test; patients who are discovered to have a TP53 mutation will be removed from study after cycle one and can continue on carfilzomib, lenalidomide, and dexamethasone (KRd); all enrolled patients will be followed for toxicity
* Subjects who have not recovered from toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of alopecia (grade 2 or 3 toxicities from prior antitumor therapy that are considered irreversible [defined as having been present and stable for > 6 months], such as grade 2 chemotherapy-induced peripheral neuropathy, may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and sponsor)
* Subjects who are receiving any other investigational agents
* Subjects who have undergone major surgery within 28 days of study day 1; vertebroplasty and/or kyphoplasty, which must have been performed at least 1 week prior to starting KRT-232 (AMG 232) + KRd
* Subjects with known central nervous system involvement of myeloma should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Subjects with history of allergic reactions attributed to compounds of similar chemical or biologic composition to KRT-232 (AMG 232) or carfilzomib, lenalidomide, or dexamethasone
* Subjects' medication list such as herbal medicines (e.g., St. John's wort), vitamins, and supplements will be reviewed before starting first dose of KRT-232 (AMG 232) and at each clinic visit; any potential drug interactions will be brought and discussed with the principal investigator; use of any known CYP3A4 substrates with narrow therapeutic window (such as alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, sirolimus, or terfanide) within the 14 days prior to receiving the first dose of KRT-232 (AMG 232) is not permitted; other medications (such as fentanyl and oxycodone) may be allowed per investigator's assessment/evaluation
* Treatment with medications known to cause QTc interval prolongation within 7 days of study day 1 is not permitted unless approved by the sponsor; use of ondansetron is permitted for treatment of nausea and vomiting
* Current use of warfarin, factor Xa inhibitors and direct thrombin inhibitors; Note: low molecular weight heparin and prophylactic low dose warfarin are permitted; PT/PTT must meet the inclusion criteria; subjects taking warfarin must have their INR followed closely
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects with myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association [NYHA] class III and higher), unstable angina, or cardiac arrhythmia requiring medication are excluded
* Subjects with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
* Subjects with history of bleeding diathesis
* Subjects with active infection requiring IV antibiotics within 2 weeks of study enrollment (day 1) are excluded
* Positive hepatitis B surface antigen (HepBsAg) (indicative of chronic hepatitis B), positive hepatitis total core antibody with negative HBsAG (suggestive of occult hepatitis B), or detectable hepatitis C virus RNA by a polymerase-chain reaction (PCR) assay (indicative of active hepatitis C - screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive); subjects with hepatitis B virus suppressed on therapy, and previously treated/eradicated hepatitis C virus are eligible for study
* Human immunodeficiency virus (HIV)-positive subjects positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive subjects must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based test
* Pregnant women are excluded from this study because KRT-232 (AMG 232) is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with KRT-232 (AMG 232), breastfeeding should be discontinued if the mother is treated with KRT-232 (AMG 232); these potential risks may also apply to other agents used in this study
* Women who are lactating/breast feeding or who plan to breastfeed while on study through 1 week after receiving the last dose of study drug
* Subjects with prior treatment with an MDM2 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Lee, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (7):
- United States (7):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Texas at Austin, Austin, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened to accrual on 10/2017 at 6 sites across ETCTN network (MD Anderson, UC Davis, UT San Antonio, UT Austin, University of Utah, Weill Cornell). Study closed to accrual 07/2024 due to uncertain development plan of MDM2 inhibitors in myeloma and slow accrual after discussion with NCI CTEP leadership and study industry collaborator, Kartos Therapeutics.
Pre-assignment Details: Accrual process was slow due to various reasons including multiple screen failures for reasons including inability to perform integral biomarker testing for TP53 mutation status due to <5% plasma cells in bone marrow biopsy at screening, TP53 mutation detected, not having measurable disease, and low creatinine clearance below eligibility threshold. 35 patients were consented, of those16 patients were eligible and dosed.
Groups:
- Part A (Dose-escalation) 60mg; Part A (Dose-escalation) 90mg; Part A (Dose-escalation) 120mg; Part A (Dose-escalation) 190mg; Part A (Dose-escalation) 240mg: Escalating doses of KRT-232 (DL1 60 mg, DL2 90 mg, DL3 120 mg, DL4 190 mg, DL5 240 mg) in combination with Carfilzomib, Lenalidomide, Dexamethasone (KRd)
- Part B (Dose-expansion): 10 patient dose-exansion at RP2D determined from Part A
Period: 60 mg
Arm/Group | Part A (Dose-escalation) 60mg | Part A (Dose-escalation) 90mg | Part A (Dose-escalation) 120mg | Part A (Dose-escalation) 190mg | Part A (Dose-escalation) 240mg | Part B (Dose-expansion)
Started | 6 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Alternative Treatment | 1 | 0 | 0 | 0 | 0 | 0
Period: 90mg
Arm/Group | Part A (Dose-escalation) 60mg | Part A (Dose-escalation) 90mg | Part A (Dose-escalation) 120mg | Part A (Dose-escalation) 190mg | Part A (Dose-escalation) 240mg | Part B (Dose-expansion)
Started | 0 | 10 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 7 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Alternative Treatment | 0 | 1 | 0 | 0 | 0 | 0
Not completed — TP53 mutation or indeterminate TP53 mutation status | 0 | 2 | 0 | 0 | 0 | 0
Period: 120mg
Arm/Group | Part A (Dose-escalation) 60mg | Part A (Dose-escalation) 90mg | Part A (Dose-escalation) 120mg | Part A (Dose-escalation) 190mg | Part A (Dose-escalation) 240mg | Part B (Dose-expansion)
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 190mg
Arm/Group | Part A (Dose-escalation) 60mg | Part A (Dose-escalation) 90mg | Part A (Dose-escalation) 120mg | Part A (Dose-escalation) 190mg | Part A (Dose-escalation) 240mg | Part B (Dose-expansion)
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 240mg
Arm/Group | Part A (Dose-escalation) 60mg | Part A (Dose-escalation) 90mg | Part A (Dose-escalation) 120mg | Part A (Dose-escalation) 190mg | Part A (Dose-escalation) 240mg | Part B (Dose-expansion)
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Relapsed and/or refractory TP53 WT Multiple Myeloma subjects with 1-3 lines of prior therapy.
Groups:
- Part A (Dose-escalation) 60 mg; Part A (Dose-escalation) 90 mg; Part A (Dose-escalation) 120 mg; Part A (Dose-escalation) 190 mg; Part A (Dose-escalation) 240 mg: Escalating doses of KRT-232 (DL1 60 mg, DL2 90 mg, DL3 120 mg, DL4 190 mg, DL5 240 mg) in combination with Carfilzomib, Lenalidomide, Dexamethasone (KRd)
- Total: Total of all reporting groups
Arm/Group | Part A (Dose-escalation) 60 mg | Part A (Dose-escalation) 90 mg | Part A (Dose-escalation) 120 mg | Part A (Dose-escalation) 190 mg | Part A (Dose-escalation) 240 mg | Total
Number analyzed (Participants) | 6 | 10 | 0 | 0 | 0 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  |  | 0
  Between 18 and 65 years | 3 | 6 |  |  |  | 9
  >=65 years | 3 | 4 |  |  |  | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 |  |  |  | 7
  Male | 3 | 6 |  |  |  | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 |  |  |  | 5
  Not Hispanic or Latino | 3 | 8 |  |  |  | 11
  Unknown or Not Reported | 0 | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  |  | 0
  Asian | 0 | 1 |  |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
  Black or African American | 0 | 2 |  |  |  | 2
  White | 4 | 6 |  |  |  | 10
  More than one race | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 2 | 1 |  |  |  | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 10 |  |  |  | 16

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Safety and Tolerability of KRT-232 (AMG 232) in Combination With Carfilzomib, Lenalidomdie, and Dexamethasone (KRd)
Time Frame: at least 6 months of treatment, an average of 1 year
Population: Only included DLT-evaluable patients. 6 of 6 patients enrolled on Dose Level 1 and 5 of 10 patients at dose level 2 were DLT-evaluable. Therefore, the primary outcome of determining the safety and tolerability beyond dose level one was not possible, and the MTD and recommended phase 2 dose could not be evaluated prior to study closure.
Measure: Number; unit: Dose Limiting Toxicity
Groups:
- Part A: Dose Level 1: KRT-232 60 mg + KRd
- Part A: Dose Level 2: KRT-232 90 mg + KRd
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 2
Number analyzed (Participants) | 6 | 5
Dose Limiting Toxicity | 1 | 1

2. Primary Outcome: Determine Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of KRT-232 (AMG 232) in Combination With Carfilzomib, Lenalidomdie, and Dexamethasone (KRd)
Time Frame: at least 6 months of treatment, an average of 1 year
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 2
Number analyzed (Participants) | 6 | 5
mg | NA — 6 of 6 patients enrolled on Dose Level 1 and 5 of 10 patients at dose level 2 were DLT-evaluable. Therefore, the primary outcome of determining the safety and tolerability beyond dose level one was not possible, and the MTD and recommended phase 2 dose could not be evaluated prior to study closure. | NA — 6 of 6 patients enrolled on Dose Level 1 and 5 of 10 patients at dose level 2 were DLT-evaluable. Therefore, the primary outcome of determining the safety and tolerability beyond dose level one was not possible, and the MTD and recommended phase 2 dose could not be evaluated prior to study closure.

3. Secondary Outcome: Evaluate PD Effects of KRT-232 (AMG 232) Through Serum MIC-1 Levels.
Time Frame: 30 days after last dose
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points.
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Assess KRT-232 (AMG 232) Exposure-response Relationships (PD, Toxicity, and Efficacy).
Time Frame: 30 days after last dose
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points.
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: At least 6 months of treatment, an average of 1 year
Description: No patients were enrolled under Part A (Dose-escalation) 120, 190 and 240 mg.
Arm/Group | Part A (Dose-escalation) 60 mg | Part A (Dose-escalation) 90 mg | Part A (Dose-escalation) 120 mg | Part A (Dose-escalation) 190 mg | Part A (Dose-escalation) 240 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/10 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/6 | 7/10 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 10/10 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Dose-escalation) 60 mg (N=6) | Part A (Dose-escalation) 90 mg (N=10) | Part A (Dose-escalation) 120 mg (N=0) | Part A (Dose-escalation) 190 mg (N=0) | Part A (Dose-escalation) 240 mg (N=0)
Eye disorders - Other, specify - Vision Decreased (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | NA | NA | NA
Infections & infestations - Other - Covid-19 Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 1 | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
White blood cell decreased (Blood and lymphatic system disorders) | 1 | 0 | NA | NA | NA
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Dose-escalation) 60 mg (N=6) | Part A (Dose-escalation) 90 mg (N=10) | Part A (Dose-escalation) 120 mg (N=0) | Part A (Dose-escalation) 190 mg (N=0) | Part A (Dose-escalation) 240 mg (N=0)
White blood cell decreased (Investigations) | 6 | 6 | NA | NA | NA
Lymphocyte count decreased (Investigations) | 5 | 6 | NA | NA | NA
Platelet count decreased (Investigations) | 6 | 4 | NA | NA | NA
Anemia (Blood and lymphatic system disorders) | 5 | 4 | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 3 | 6 | NA | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 4 | NA | NA | NA
Neutrophil count decreased (Investigations) | 6 | 3 | NA | NA | NA
Fatigue (General disorders) | 2 | 6 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 2 | 6 | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3 | NA | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3 | NA | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 3 | NA | NA | NA
Insomnia (Psychiatric disorders) | 2 | 4 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 2 | 3 | NA | NA | NA
Headache (Nervous system disorders) | 2 | 3 | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 2 | 3 | NA | NA | NA
Alkaline phosphatase increased (Investigations) | 2 | 2 | NA | NA | NA
Creatinine increased (Investigations) | 1 | 3 | NA | NA | NA
Edema limbs (General disorders) | 2 | 2 | NA | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1 | NA | NA | NA
ALT increased (Investigations) | 1 | 2 | NA | NA | NA
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | NA | NA | NA
Chills (General disorders) | 1 | 2 | NA | NA | NA
Dizziness (Nervous system disorders) | 2 | 1 | NA | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | NA | NA | NA
Fever (General disorders) | 1 | 2 | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | NA | NA | NA
Investigations - Other, specify - Blood Bicarbonate Decreased (Investigations) | 1 | 2 | NA | NA | NA
Investigations - Other, specify - Ldh Increased (Investigations) | 1 | 2 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | NA | NA | NA
AST increased (Investigations) | 1 | 1 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 | 1 | NA | NA | NA
Bruising (Skin and subcutaneous tissue disorders) | 2 | 0 | NA | NA | NA
Cataract (General disorders) | 1 | 1 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA | NA
Cystitis noninfective (Renal and urinary disorders) | 2 | 0 | NA | NA | NA
Dysgeusia (Nervous system disorders) | 1 | 1 | NA | NA | NA
Hematuria (Renal and urinary disorders) | 1 | 1 | NA | NA | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | NA | NA | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 1 | NA | NA | NA
Investigations - Other, specify - Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 2 | NA | NA | NA
Investigations - Other, specify - Hyperphosphatemia (Investigations) | 2 | 0 | NA | NA | NA
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 2 | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | NA | NA | NA
Proteinuria (Renal and urinary disorders) | 1 | 1 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | NA | NA | NA
Superficial thrombophlebitis (Vascular disorders) | 1 | 1 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 1 | NA | NA | NA
AV block first degree (Cardiac disorders) | 0 | 1 | NA | NA | NA
Anxiety (General disorders) | 0 | 1 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 1 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA
Cardiac troponin T increased (Investigations) | 0 | 1 | NA | NA | NA
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA
Dry eye (General disorders) | 0 | 1 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA
EKG QT corrected interval prolong (Investigations) | 0 | 1 | NA | NA | NA
Ejection fraction decreased (Investigations) | 1 | 0 | NA | NA | NA
Endocarditis infective (Infections and infestations) | 0 | 1 | NA | NA | NA
Enterocolitis infectious (Infections and infestations) | 0 | 1 | NA | NA | NA
Eye disorders - Other, specify - Blurred Vision Bilateral (General disorders) | 0 | 1 | NA | NA | NA
Eye disorders - Other, specify - Left Eye Stye (General disorders) | 0 | 1 | NA | NA | NA
Floaters (General disorders) | 1 | 0 | NA | NA | NA
Flushing (General disorders) | 1 | 0 | NA | NA | NA
GGT increased (Investigations) | 1 | 0 | NA | NA | NA
Gait disturbance (General disorders) | 0 | 1 | NA | NA | NA
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | NA | NA | NA
Infections & infestations - Other - Shingles (Infections and infestations) | 0 | 1 | NA | NA | NA
Infections & infestations - Other - Viral Infections Nos (Infections and infestations) | 0 | 1 | NA | NA | NA
Infusion related reaction (General disorders) | 1 | 0 | NA | NA | NA
Investigations - Other, specify - Bbc Decreased (Investigations) | 0 | 1 | NA | NA | NA
Investigations - Other, specify - Total Protein Decreased (Investigations) | 0 | 1 | NA | NA | NA
Investigations - Other, specify - Total Protein Increased (Investigations) | 0 | 1 | NA | NA | NA
Irritability (General disorders) | 1 | 0 | NA | NA | NA
Libido decreased (General disorders) | 1 | 0 | NA | NA | NA
Memory impairment (Nervous system disorders) | 1 | 0 | NA | NA | NA
Metabolism and nutrition - Other - Blood Bicarbonate Decreased (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA
Metabolism and nutrition - Other - Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA
Musculoskel/connect tissue -Other - Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA | NA
Musculoskel/connect tissue -Other - Muscle Cramps - Hands (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA | NA
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA
Oral pain (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA
Pain (General disorders) | 1 | 0 | NA | NA | NA
Palpitations (Cardiac disorders) | 1 | 0 | NA | NA | NA
Toothache (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA | NA
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA | NA
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA
Reproductive and breast - Other - Vaginal Itching (General disorders) | 1 | 0 | NA | NA | NA
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 1 | 0 | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 1 | NA | NA | NA
Skin & subcutaneous tissue -Other - Facial Tightening (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA
Skin infection (Infections and infestations) | 1 | 0 | NA | NA | NA
Tremor (Nervous system disorders) | 0 | 1 | NA | NA | NA
Upper respiratory infection (Infections and infestations) | 1 | 0 | NA | NA | NA
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | NA | NA | NA
Vaginal infection (Infections and infestations) | 0 | 1 | NA | NA | NA
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03031730/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03031730/ICF_001.pdf